CLINICAL TRIAL: NCT05172232
Title: A Prospective Clinical Investigation to Assess the Diagnostic Precision of the AI Tool Dermalyzer to Identify Malignant Melanomas in Subjects Seeking Primary Care for Melanoma-suspected Cutaneous Lesions
Brief Title: Diagnostic Precision of the AI Tool Dermalyzer to Identify Malignant Melanomas in Subjects Seeking Primary Care for Melanoma-suspected Cutaneous Lesions
Acronym: AI-DSMM
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Collaborators: Karolinska Institutet (Other); Region Östergötland (Other); Region Stockholm (Other Government); Landstinget i Kalmar Län (Other); Kronoberg County Council (Other Government)
Responsible Party: Principal Investigator, Magnus Falk, Associate professor, Linkoeping University
Other Study IDs: CIV-21-12-038346
Record Dates: First submitted 2021-12-23; First posted 2021-12-29 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Malignant Melanoma
Keywords: artificial intelligence; diagnostic accuracy; clinical desicion supportive tool
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary care patients with melanoma suspicious skin lesion(s): Patients seeking primary care, having one or more skin lesion that the primary care physician cannot by certainty can rule out as being a possible melanoma.
  Interventions: Diagnostic Test: Dermalyzer

INTERVENTIONS:
Diagnostic Test: Dermalyzer — To evaluate the diagnostic accuracy of the Dermalyzer device to detect melanoma among cutaneos skin lesions by dermoscopy.

SUMMARY:
Dermalyzer is a device intended to be used as a decision support system for assessing cutaneous lesions suspected of being melanomas. The input from the device is not intended to be used as the sole source of information for diagnosis. Intended to be used by medical professionals. The service does not provide any other diagnosis. The study is a pre-marketing, prospective, confirmatory, first in clinical setting, pivotal multi-centre, non-interventional clinical investigation to evaluate the clinical safety, performance and benefit of Dermalyzer in patients with cutaneous lesions where malignant melanoma (MM) cannot be ruled out.

Primary objective: The primary objective of the investigation is to determine the diagnostic precision of the device; to answer at which level the AI tool Dermalyzer can identify malignant melanomas among cutaneous lesions that are assessed in clinical use due to any degree of malignancy suspicion.

Secondary objectives: A) To evaluate usability and applicability in clinical praxis of Dermalyzer by users (medical professionals), B)To gain an increased knowledge and understanding of how digital tools enhanced co-artificial intelligence can assist physicians with the right support for an earlier diagnosis of malignant melanoma.

Exploratory objective: To explore health economic aspects of improved diagnosis support

Methods: The subjects will be included from around 30 primary care centers in Sweden. If the subject's lesion(s) is suspected of melanoma or melanoma cannot be ruled out, the subject is asked to participate in the investigation. The investigator examines the subject's lesion(s) and makes the clinical assessment of the subject lesion(s) based on established clinical decision algorithms The investigator takes dermoscopy images according to standard of care and archives the image(s) according to clinical routine. The investigator decides on action, based on his or her MM suspicion (excision at the primary care center or referral for excision or referral to a dermatologist for further assessment). The investigator takes images of the lesion(s) again, this time with a mobile phone, containing the AI software, connected to a dermatoscope, and follows the on-screen instructions. The image is processed by the AI and the results are visible on the screen within seconds. The investigator records how he considers that the degree of suspicion of MM (higher vs lower) would have been affected by the AI SW result if it had been the governing body for the treatment. At study follow-up, the final tumor diagnosis from the histopathology results (melanoma/non melanoma) or by dermatologist assessment (if stated as undoubtedly benign), the degree of agreement between the true final diagmosis and the outcome of the AI decision support is determined, and the diagnostic accuracy in distinguishing melanoma from non-melanoma, in terms of sensitivity and specificity as well the positive and predictive value. The corresponding comparison is performed from the examining investigators estimated clinical degree of suspicion. The clinical investigation will collect information from the users, how participating users (investigators at the site) experience the usability of the AI decision support and attaching applications, from short surveys including the validated System Usability Scale.

DETAILED DESCRIPTION:
Background: Malignant melanoma is a worldwide health issue of concern, of increasing incidence. Early melanoma detection is crucial for survival and prognosis. Dermalyzer is a device intended to be used as a decision support system for assessing cutaneous lesions suspected of being melanomas, based on artificial intelligence (AI), often referred to as "machine learning". The input from the device is not intended to be used as the sole source of information for diagnosis. Intended to be used by medical professionals. The service does not provide any other diagnosis.

Study aims/objectives:

Primary objective: The primary objective of the investigation is to determine the diagnostic precision of the device; to answer at which level the AI tool Dermalyzer can identify malignant melanomas among cutaneous lesions that are assessed in clinical use due to any degree of malignancy suspicion.

Secondary objectives: A) To evaluate usability and applicability in clinical praxis of Dermalyzer by users (medical professionals), and B) To gain an increased knowledge and understanding of how digital tools enhanced co-artificial intelligence can assist physicians with the right support for an earlier diagnosis of malignant melanoma.

Exploratory objective: To explore health economic aspects of improved diagnosis support Exploratory endpoints

Materials & methods:

The subjects will be included from around 30 primary care centers in Sweden. If the subject's lesion(s) is suspected of melanoma or melanoma cannot be ruled out, the subject is asked to participate in the investigation. The investigator examines the subject's lesion(s) and makes the clinical assessment of the subject lesion(s) based on established clinical decision algorithms (such as "Chaos & clues", "3- or 7-point checklist", or the ABCDE concept) of whether there is a suspicion of MM, according to the usual clinical routine (also includes very low suspicion of MM but cannot be completely dismissed). The investigator takes dermoscopy images according to standard of care and archives the image(s) according to clinical routine. The investigator decides on action, based on his or her MM suspicion (excision at the primary care center or referral for excision or referral to a dermatologist for further assessment). If the subject has agreed to participate in the investigation, the investigator indicates in the CRF the clinical suspicion level of MM, and decided action. The investigator takes images of the lesion(s) again, this time with a mobile phone, containing the IMD AI SW, connected to a dermatoscope, and follows the on-screen instructions. The image is processed by the AI SW and the results are visible on the screen within seconds. A unique auto generated code number is also presented. The code number is registered on the enrollment log and in the CRF. The investigator records how he considers that the degree of suspicion of MM (higher vs lower) would have been affected by the AI SW result if it had been the governing body for the treatment.

When the subject has been fully examined and receives the final tumor diagnosis from the histopathology/PAD results or dermatologist assessment (melanoma/non melanoma), the degree of agreement between the PAD and the outcome of the AI SW decision support is calculated with the Kappa-analysis and the diagnostic accuracy to be able to distinguish melanoma from non-melanoma in the form of sensitivity and specificity as well the positive and predictive value. The corresponding comparison is performed from the examining investigators estimated clinical degree of suspicion, as well as the diagnostic accuracy when both the PAD and the AI decision support are wigheted together (ei in cases where the investigator and the decisions support are in agreement in their assessment). The clinical investigation will collect information from the users, how participating users (investigators at the site) experience the usability of the AI SW decision support and attaching applications, from short surveys including the validated System Usability Scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years
* Patients attending a primary care facility with at least 1 suspicious skin lesion where malignant melanoma cannot be ruled out.
* Willingness and ability to provide informed consent.

Exclusion Criteria:

* Cutaneous lesions that are considered as benign by the investigator and thus not subject for further clinical investigation
* Cutaneous lesions in areas that are not suitable for dermoscopy imaging
* Cutaneous lesions in areas with any form of scarring of tissue due to injury
* Damaged or injured non intact skin where the cutaneous lesion is located
* Individuals with skin type V and VI according to the Fitzpatrick scale (darker brown or black coloured skin)
* Cutaneous lesions in areas covered by tattoos
* Cutaneous lesions in abundantly hairy skin areas (provided the the area cannot be shaved freely from the hair to allow clear view for the dermatoscope)
* Images where the entire lesion is not inside the photo
* Images that are out of focus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care patients
Sampling Method: Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Falk, Ass.Prof., Principal Investigator — Linkoeping University
Locations (3):
- Sweden (3):
  - Region Östergötland Primary Care, Linköping, Docent
  - Region Stockholm Primary Care, Stockholm
  - Region Kalmar and Kronoberg, Vaxjo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Care Patients With Melanoma Suspicious Skin Lesion(s)
Started | 231
Completed | 228
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Primary Care Patients With Melanoma Suspicious Skin Lesion(s)
Number analyzed (Participants) | 228
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [55 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125
  Male | 103
Race/Ethnicity, Customized [Number; unit: participants] — Fitzpatrick's Skin type
  participants
    Skin type 1: Pale skin, easily burns, never tans, often blond or red hair (assessed by physician) | 19
    Skin type 2: Fair skin, easily burns, seldom tans (assessed by physician) | 145
    Skin type 3: Darker white skin, sometimes burns, easily tans (assessed by physician) | 52
    Skin type 4: Light brown skin, seldom burns, always tans (assessed by physician) | 12
Region of Enrollment [Number; unit: participants]
  Sweden | 228
Clinical suspicion degree of melanoma (asssessed by examining physician) [Count of Participants; unit: Participants]
  Low degree of suspicion, but cannot exclude melanoma. | 177
  High degree of suspicion of melanoma | 51

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy to Detect Melanoma
Description: The number of correctly classified skin lesions by the Dermalyzer (melanoma vs not melanoma), as compared with the result of the standard diagnostic procedure (dermatologist assessment and histoptahologic analysis).
Time Frame: 12 months
Population: Patients with some degree ov melanoma suspsicion raised by the examining primary care physician.
Measure: Number; unit: number of skin lesions
Units Other Than Participants: uniqe skin lesions
Groups:
- Diagnostic Accuracy of Dermalyzer to Detect Melanoma: Proportions of melanoma and non-melanoma skin lesions identified by Dermalyser, as compared to the true diagnosis set by the conventional, standard diagnostic procedure.
Arm/Group | Diagnostic Accuracy of Dermalyzer to Detect Melanoma
Number analyzed (Participants) | 228
Number analyzed (uniqe skin lesions) | 253
number of skin lesions
  True positives | 20
  False positives | 92
  False negatives | 1
  True negatives | 140

2. Secondary Outcome: Instrument Usability of the Device
Description: User experience and perception of the Dermalyzer, in the form of System Usability Scale, to evaluate the usability and applicability in clinical praxis. The validated scale conists of 10 Likert scale based questions (scored 1-5 points), reflecting different aspects of usability, such as easiness to use, complexity, inconsistensy, understandability, etc. It summurizes in a score ranging from 0 - 100 points, where a high score reflects good usability properties.
Time Frame: Secondary measurement variable data was collected after baseline primary data inclusion was ended in Feb 2022, and completeted within 3 months from that.
Population: Primary care physicians that took part in the recruitment and inclusion of patients (study participants) in the trial.
Measure: Median (Full Range); unit: SUS score points
Groups:
- Perceived Device Usability: System Usability Scale score
Arm/Group | Perceived Device Usability
Number analyzed (Participants) | 138
SUS score points | 75 [47.5 to 87.5]

ADVERSE EVENTS:
Time Frame: Possible adverse events were collected during the single patient visit at which the patients (participants) were exposed to the device tested (the Dermalyzer). Approximately, such a visit took 15-20 minutes, and also checked att the time of retreiving the skin lesion diagnosis from the patient record.
Arm/Group | Primary Care Patients With Melanoma Suspicious Skin Lesion(s)
All-Cause Mortality (participants affected / at risk) | 0/231
Serious Adverse Events (participants affected / at risk) | 0/231
Other Adverse Events (participants affected / at risk) | 0/231

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT05172232/Prot_SAP_000.pdf